CLINICAL TRIAL: NCT01581190
Title: Comparison of Bananas and Gatorade on Performance and Exercise-induced Inflammation, Oxidative Stress, and Changes in Immune Function in Endurance Athletes
Brief Title: Bananas as an Energy Source During Exercise: a Metabolomics Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: Dole Food Company (Industry)
Responsible Party: Principal Investigator, David C. Nieman, Professor, Director of the Human Performance Lab, Appalachian State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-0082
Record Dates: First submitted 2012-04-14; First posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Intense Exercise
Keywords: Bananas; Exercise; Metabolomics; Oxidative stress; Inflammation; Immune function
MeSH Terms: conditions — Motor Activity; Inflammation | interventions — gatorade

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bananas versus 6% carbohydrate beverage (Experimental)
  Interventions: Dietary Supplement: Bananas versus 6% carbohydrate beverage

INTERVENTIONS:
Dietary Supplement: Bananas versus 6% carbohydrate beverage — Trained cyclists (N=14) completed two 75-km cycling time trials (randomized, crossover) while ingesting BAN or CHO (0.2 g/kg carbohydrate every 15 min).
  Other Names: Gatorade

SUMMARY:
This study compared the acute effect of ingesting bananas (BAN) versus a 6% carbohydrate drink (CHO) on 75-km cycling performance and post-exercise inflammation, oxidative stress, and innate immune function using traditional and metabolomics-based profiling.

DETAILED DESCRIPTION:
Trained cyclists (N=14) completed two 75-km cycling time trials (randomized, crossover) while ingesting BAN or CHO (0.2 g/kg carbohydrate every 15 min). Pre-, post-, and 1-h-post-exercise blood samples were analyzed for glucose, granulocyte (GR) and monocyte (MO) phagocytosis (PHAG) and oxidative burst activity, nine cytokines, F2-isoprostanes, ferric reducing ability of plasma (FRAP), and metabolic profiles using gas chromatography-mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Ages 18-45 years
* Cyclists, road racing experience.
* Willing to avoid the use of supplements, herbs, medications during the study.

Exclusion Criteria:

* Female
* Over the age of 45 years
* No cycling racing experience
* Using supplements and medications during the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Performance and fuel substrate utilization as measured through metabolomics | Up to 6 months
  Will measure shifts in metabolites following 75-km cycling while ingesting bananas or 6% carbohydrate beverage. The shift in metabolites will be assessed using GC-MS. Time frame from date of randomization until the last samples are collected and analyzed will be up to six months.

SECONDARY OUTCOMES:
Exercise-induced inflammation. | up to 6 months
  Cytokine panel (IL-6, IL-8, IL-10, TNF-alpha) before and after cycling 75-km; measured with Meso Scale Discovery in pg/ml. Time frame from randomization until the last samples are collected and analyzed will be up to six months.

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State University
Locations (1):
- Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

REFERENCES:
- See also: Website for lab — http://www.ncrc.appstate.edu